CLINICAL TRIAL: NCT07242287
Title: Comparison of15-Minute Home-Based Flexibility Exercises Derived by Artificial Intelligence and Produced by Humans on the Overall Flexibility, Back Health, and Muscle Stiffness Levels of Office Workers: A Randomized Controlled Trial
Brief Title: Flexibility Exercises, Created by AI and Humans, on Office Workers' Flexibility, Back-health and Muscle-stiffness.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Mehmet Sönmez, Assistant Doctor, Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mehmet.sonmez2
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Office Workers
Keywords: Flexibility exercises; AI-created; Human-created; Muscle stiffness; back health; flexibility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15-Minute Home-Based Flexibility Exercises Derived by Artificial Intelligence Group (Experimental): An AI-powered platform called Gemini will automatically generate a standardized 15-minute flexibility exercise program for each participant. This program will include dynamic and static stretching exercises.
  Interventions: Other: AI-created exercise
- 15-Minute Home-Based Flexibility Exercises Producted by Human Group (Experimental): For this group, a 15-minute program consisting of standardized flexibility exercises modified for each participant based on calisthenic exercises (bodyweight exercises) will be created by two qualified physical therapists. This program will target similar muscle groups and have the same duration as the AI group's program.
  Interventions: Other: Human-created exercise

INTERVENTIONS:
Other: AI-created exercise — 15-minute home flexibility exercise program derived by artificial intelligence over 4 weeks
  Other Names: Flexibility exercise derived by AI
  Arms: 15-Minute Home-Based Flexibility Exercises Derived by Artificial Intelligence Group
Other: Human-created exercise — 15-minute home flexibility exercise program producted by human over 4 weeks
  Other Names: Flexibility exercises producted by human
  Arms: 15-Minute Home-Based Flexibility Exercises Producted by Human Group

SUMMARY:
While the benefits of flexibility exercises for office workers are well known, there is no randomized controlled comparison to determine whether these exercises can be delivered more effectively and safely by a specialist or by an automated artificial intelligence algorithm. Furthermore, considering the dynamic programming potential of artificial intelligence, determining whether this method can provide results similar to or superior to traditional methods is critical for the development of future healthcare models. The primary objective of this study is to compare the effects of 15-minute home-based flexibility exercises derived by artificial intelligence and produced by humans, administered over a 4-week period, on office workers' overall flexibility, back health, and muscle stiffness levels. This study is a two-armed, single-blind randomized controlled trial. Participants will be blinded to which group they are assigned to. This study will be respond "Are flexibility exercises generated by artificial intelligence more effective than human-generated flexibility exercises" question. During the study, participants who sign the volunteer information form and consent form and meet the inclusion criteria will be divided equally into two groups using a simple random method (coin toss):

* Group A: Artificial Intelligence (AI)-Based Flexibility Group.
* Group B: Human Expert-Based Flexibility Group. Intervention programs will include a standardized 15-minute flexibility exercise program will be automatically generated for each participant via Gemini, an AI-powered platform for group A, and a 15-minute program consisting of standardized flexibility exercises modified for each participant created by two qualified physiotherapists, based on calisthenic exercises (using body weight). This program will target the same muscle groups as the AI group's program and will be of similar duration. The exercise program will last a total of 4 weeks. Participants will exercise 3 days a week (Monday, Wednesday, Friday) for 15 minutes a day in their own environment.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial. The hypothesis of the study;

* HO1: Flexibility exercises generated by artificial intelligence improve overall flexibility in office workers more than human-generated flexibility exercises.
* HO2: Flexibility exercises generated by artificial intelligence reduce back pain levels in office workers more than human-generated flexibility exercises.
* HO3: Flexibility exercises generated by artificial intelligence are more effective than human-generated flexibility exercises in relaxing muscle stiffness in office workers.

Office workers employed at Erzurum Technical University will be included in the study. The minimum number of participants required for the study was determined to be 21 people per group using the Gpower 3.1 (Düsseldorf, Germany) program, with a 0.05 margin of error, 95% confidence interval, and 1.03 effect size.

All participants' pre-test (baseline) and post-test measurements at the end of the 4-week intervention period will be collected under the same conditions and in the same environment. The exercises for both groups will be provided to them as a brochure after the first measurement session, and instructions on how to perform them will be given. The intervention period will last for 4 weeks. On exercise days-Monday, Wednesday, and Friday-participants will receive reminder messages via the designated online communication group to remind them to do their exercises. Participants will be asked to provide brief feedback confirming they have completed the exercises for compliance tracking.

The AI-generated flexibility exercises will consist of a 2-minute warm-up, 11 minutes of stretching and flexibility exercises (including static and dynamic stretches), and a 2-minute cool-down. Human-generated flexibility exercises will consist of a 2-minute warm-up modified from calisthenic exercises, 11 minutes of main flexibility exercises (squats, modified push-ups, planks, etc.), and a 2-minute cool-down.

In our study, a demographic data collection form will be used to evaluate demographic data, the sit-and-reach test for flexibility assessment, the Oswestry Disability Index to assess back health, and the MyotonPRO muscle tone assessment device to evaluate muscle stiffness.

All measurements will be conducted in two sessions at the Therapeutic Exercise Laboratory of Erzurum Technical University. Measurements will be taken immediately before the start of the study and after the 4-week training period. An informed consent form will be obtained from each participant, and the test procedures will be explained in detail. Measurements will be performed by an experienced physical therapist in accordance with standardized protocols. Participants will be given sufficient rest time before each test, and their safety will be ensured. The total assessment time is estimated to be 12 minutes for each participant.

The obtained data will be analyzed using the SPSS 24.0 (Statistical Package for the Social Sciences) program. At the same time, comparisons will be made by entering the norm values into the SPSS 24.0 program. The Kolmogorov-Smirnov or Shapiro-Wilk tests will be used to examine whether the data are normally distributed. Descriptive statistics (mean, standard deviation) will be used for normally distributed data. The X2 test will be used for categorical variables. The independent samples t-test will be used to compare independent groups. Non-parametric tests (e.g., Mann-Whitney U test) will be preferred for data that do not show a normal distribution. For intra-group comparisons, the paired t-test or Wilcoxon signed rank test will be used depending on the normal distribution status of the data. In all statistical analyses, the significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Not have any known chronic orthopedic problems (active injuries requiring surgery or causing limited mobility).
* Be able to walk distances of 150 meters or more without assistance.
* Be an office worker who spends most of their working hours at a desk (at least 30 hours per week).

Exclusion Criteria:

* Having a chronic illness (cardiovascular disease, respiratory disease, metabolic disease, etc.).
* Having a condition that causes acute or chronic pain related to the musculoskeletal system.
* Having undergone major surgery within the last 6 months.
* Experiencing a health problem during participation that would cause any physical activity restrictions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Body flexibility | The change from baseline sit and reach test score at week 4.
  The sit-and-reach test will be used for evaluation. This test measures body flexibility and is performed on a specially developed sit-and-reach bench. Sit with both legs straight on the floor. One hand is placed on top of the other with the middle fingertips aligned. The soles of the feet are placed on the footrest of the measuring device. The subject is instructed to inhale and then, while exhaling, bend at the hips and reach forward, pushing the sliding ruler on the device. The back should be straight and the head up. Avoid jumping or rapid movements, and never stretch to the point of pain. Keep the knees straight and hold the reaching position for 2 seconds. Record the distance traveled by the sliding ruler in centimeters. Perform two trials. Record the longest distance. This is a valid and safe test.
Back health | The change from baseline Oswestry Disability Index score at week 4.
  It will be assessed using the Oswestry Disability Index. This questionnaire, which assesses back health in 10 categories, is calculated out of a total of 50 points. A high score indicates a poor prognosis.
Muscle stiffness | The change from baseline MyotonPRO device score at week 4.
  The MyotonPRO muscle characteristics assessment device will be used for evaluation. This device provides the ability to measure changes in muscle tone instantly and objectively. It has been developed to assess muscle tone, muscle stiffness, and muscle elasticity. It is a reliable measurement device for assessing back health. The assessment will be performed on the muscle groups most related to back health and flexibility limitations in office workers, namely the lumbar erector spinae (lower back), hamstrings (back of the thigh), and gastrocnemius medialis (calf).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet SÖNMEZ, PhD, Study Chair — Erzurum Technical University
Locations (1):
- Erzurum Technical University Health Science Faculty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No